CLINICAL TRIAL: NCT02503462
Title: Effect of Cobicistat Versus Ritonavir Boosting on the Brain Permeation of Darunavir in HIV-infected Individuals
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: No additional patients fulfilling the inclusion criteria
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DRVCOBI
Record Dates: First submitted 2015-07-09; First posted 2015-07-21 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: AIDS-related Dementia Complex
Keywords: HIV; darunavir; ritonavir; cobicistat; CSF; pharmacokinetics
MeSH Terms: conditions — AIDS Dementia Complex | interventions — Darunavir; Ritonavir; Cobicistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- darunavir/ritonavir vs cobicistat (Experimental): All HIV infected patients will be treated with a darunavir/ritonavir (800/100 mg) once daily containing regimen. Darunavir/ritonavir concentrations will be measured simultaneously in CSF and plasma after 1 month of treatment. The treatment will be switched to darunavir/cobicistat (800/150 mg) once daily and darunavir/cobicistat levels will be measured in CSF and plasma after 1 month of treatment.
  Interventions: Drug: Darunavir; Drug: ritonavir; Drug: cobicistat

INTERVENTIONS:
Drug: Darunavir — darunavir 800 mg once daily will be first given together with ritonavir 100 mg once daily for one month (period 1) and then darunavir 800 mg once daily will be given together with cobicistat 150 mg once daily for one month (period 2). Afterwards, all patients will be switched back to darunavir/ritonavir (800/100 mg once daily).
  Other Names: Prezista
Drug: ritonavir — ritonavir 100 mg once daily will be used to boost darunavir 800 mg once daily (period 1).
  Other Names: Norvir
Drug: cobicistat — cobicistat 150 mg once daily will be used to boost darunavir 800 mg once daily (period 2).
  Other Names: Tybost

SUMMARY:
The purpose of this study is to assess whether a boosting by cobicistat results in similar concentrations of darunavir in the brain compared to a boosting by ritonavir.

DETAILED DESCRIPTION:
Cobicistat is a new pharmacokinetic enhancer or booster of the HIV protease inhibitor darunavir. Cobicistat is distinct from the conventional booster ritonavir in that cobicistat presents a more selective inhibition of the enzymes metabolizing drugs. In addition, cobicistat is a weaker inhibitor of the efflux drug transporters expressed at the level of the blood-brain barrier (i.e. P-glycoprotein (P-gp) and breast cancer resistance Protein (BCRP)). A weaker inhibition of these efflux transporters could possibly result in less darunavir entering the brain when boosted by cobicistat as compared to a boosting by ritonavir. Such a difference could potentially be critical in patients with HIV-associated neurocognitive disorders as sufficient drug levels are needed to efficiently inhibit HIV replication inside the brain.

The aim of this study is to determine whether the boosting of darunavir by cobicistat results effectively in lower darunavir concentrations in the CSF as compared to a boosting by ritonavir. The study will be performed in HIV infected patients presenting HIV associated neurocognitive disorders (HAND) and requiring a lumbar puncture for clinical reasons. In addition, the patients will be only eligible if the are treated or if they qualify for a darunavir/ritonavir (800/100 mg once daily) containing regimen. Darunavir concentrations will be measured simultaneously in the CSF and plasma (CSF/plasma ratio) first with the ritonavir boosting and subsequently with the cobicistat boosting.

ELIGIBILITY:
Inclusion Criteria:

* documented HIV infection
* presence of HIV associated neurocognitive disorders requiring a lumbar puncture for clinical reasons
* treatment or qualifying to be treated with a HIV therapy including darunavir/r (800/100 mg once daily)
* ability to comply with the study requirements
* informed consent

Exclusion Criteria:

* conditions which disrupt the blood-brain barrier and thereby impact the entry of drugs in the brain (meningitis, meningoencephalitis, multiple sclerosis, progressive multifocal leucoencephalopathy)
* co-medications inhibiting/inducing P-glycoprotein and BCRP
* co-medications inhibiting/inducing cytochrome P450 isoenzyme 3A4 (CYP3A4)
* non adherence to Treatment
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-07; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Cerebrospinal fluid/plasma concentrations (ng/ml) of darunavir/ritonavir versus darunavir/cobicistat | 1 month
  darunavir concentrations (ng/ml) in the cerebrospinal fluid when coadministered with ritonavir versus cobicistat relative to the corresponding concentrations of darunavir in the plasma

SECONDARY OUTCOMES:
Cerebrospinal fluid concentrations (ng/ml) of darunavir/ritonavir versus darunavir/cobicistat relative to the concentration of darunavir (ng/ml) inhibiting 50% (IC50) or 90% (IC90) of the viral replication | 1 month
  darunavir concentrations (ng/ml) in the cerebrospinal fluid when coadministered with ritonavir versus cobicistat relative to darunavir concentrations (ng/ml) suppressing HIV replication by 50% and 90% (IC50 and IC90)
Proportion of responders (HIV RNA < 50 copies/ml in CSF) for darunavir/ritonavir versus darunavir/cobicistat | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Battegay, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Division of Infectious Diseases, University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Bartels H, Decosterd L, Battegay M, Marzolini C. Darunavir concentrations in CSF of HIV-infected individuals when boosted with cobicistat versus ritonavir. J Antimicrob Chemother. 2017 Sep 1;72(9):2574-2577. doi: 10.1093/jac/dkx165. PMID 28575323